CLINICAL TRIAL: NCT05456854
Title: Evaluation of Kisspeptin Stimulated Insulin Secretion With Hyperglycemic Clamp
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Futility
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Stephanie B. Seminara, MD, Chief, Reproductive Endocrine Unit; Professor of Medicine, Harvard Medical School; Director, Harvard Reproductive Endocrine Sciences Center, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 267335
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Metabolic Disease
MeSH Terms: conditions — Metabolic Diseases | interventions — KISS1 protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Kisspeptin (Experimental): Intravenous administration of kisspeptin 112-121 x 16 hours
  Interventions: Diagnostic Test: Hyperglycemic Clamp; Drug: Kisspeptin-10
- Placebo (Placebo Comparator): Intravenous administration of placebo x 16 hours
  Interventions: Diagnostic Test: Hyperglycemic Clamp; Drug: Placebo

INTERVENTIONS:
Diagnostic Test: Hyperglycemic Clamp — Administration of a hyperglycemic clamp
Drug: Kisspeptin-10 — Administration of kisspeptin-10 * 16 hr
  Arms: Kisspeptin
Drug: Placebo — Administration of placebo *16 hr
  Arms: Placebo

SUMMARY:
The goal of this study is to understand how exogenous kisspeptin affects metabolism by evaluating responses to an hyperglycemic clamp

DETAILED DESCRIPTION:
Assignment: Each study subject will serve as their own control. The order of the visits will be randomized.

Delivery of Interventions:

Prior to the study visit, subjects will undergo a review of their medical history and screening laboratories.

During the inpatient study, the subjects will

Undergo a 16-hour kisspeptin infusion Undergo a hyperglycemic clamp

ELIGIBILITY:
* over the age of 17
* normal pubertal development
* regular menstrual cycles
* stable weight for previous three months
* normal body mass index
* blood pressure systolic BP < 140 mm Hg, diastolic < 90 mm Hg
* normal hemoglobin
* hemoglobin A1C < 6.5%
* BUN, creatinine not elevated
* AST, ALT < 3x upper limit of normal
* negative serum pregnancy test

Exclusion Criteria:

* active illicit drug use,
* history of a medication reaction requiring emergency medical care,
* difficulty with blood draws.
* history of hypertension, diabetes, heart disease, high cholesterol, cancer, or clotting disorders.
* history of chronic disease that has required hospitalization
* recent use of prescription medications which interfere with metabolism or reproduction (recent = within 5 half-lives of the drug) unless it is birth control
* history of diabetes in a first degree relative
* hyperlipidemia by fasting lipid panel

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
First Phase Insulin Secretion | 10 minutes
  Average Change in First Phase Insulin Secretion Between Kisspeptin and Placebo Arms
Second Phase Insulin Secretion | 2 hours
  Average Change in Second Phase Insulin Secretion Between Kisspeptin and Placebo Arms

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Lippincott, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No